CLINICAL TRIAL: NCT04331938
Title: The Efficacy of Landmark-guided Percutaneous Sphenopalatine Ganglion Block on Self-reported Headache Pain Secondary to Aneurysmal Subarachnoid Hemorrhage: A Feasibility Study
Brief Title: Efficacy of Percutaneous SPG Block in Aneurysmal SAH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Narayan R. Kissoon, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-008846
Record Dates: First submitted 2020-03-27; First posted 2020-04-02 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Subarachnoid Hemorrhage; Headache
Keywords: sphenopalatine ganglion block
MeSH Terms: conditions — Subarachnoid Hemorrhage; Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label Arm (Experimental): Patients will receive a 5mL injection comprised of 4.5mL 1% bupivacaine and 0.5mL of dexamethasone (10mg/mL) directed towards the sphenopalatine ganglion. This will be performed on both sides. Patients will be asked to rate their pain pre- and 30 minutes post-procedure on a scale of 0-10. Patients will also be asked to rate their nausea and photophobia on a similar scale. Patients will be reevaluated at 24 hours and 48 hours post procedure.
  Interventions: Drug: Regional anesthetic SPG block-bilateral

INTERVENTIONS:
Drug: Regional anesthetic SPG block-bilateral — Patients will receive a 5mL injection comprised of 4.5mL 1% bupivacaine and 0.5mL of dexamethasone (10mg/mL) directed towards the sphenopalatine ganglion on each side (5 mL on each side)

SUMMARY:
Researchers are trying to develop alternative means to help patients with headache pain secondary to aneurysmal subarachnoid hemorrhage (bleeding about the brain).

DETAILED DESCRIPTION:
This study is an open label, feasibility study that will consist of fifteen patients. This study will enroll only patients who have aneurysmal SAH that are secured by endovascular coiling. When a patient notes a severe headache which requires medical intervention on at least day 3 of the hospital admission, they will be asked if they would like to participate in an open label trial to use a bilateral SSPGB in addition to traditional medical management per unit protocol. The risks and benefits of the procedure will be explained to the patient. The patient will then either agree or disagree. If the patient disagrees, they will not be enrolled in the study. If the patient agrees, they will sign an informed consent and will be enrolled. Inclusion and exclusion criteria will be reviewed before enrolling a patient. The patients will first rate their pain from 0-10 on the numeric rating scale (NRS) (10 being the most severe). If their pain is at a level 5 or more and it is not responsive to traditional medical therapies, they will be a candidate for the study. The patients will receive bilateral injections as outlined below (5 mL: 4.5mL of 0.5% bupivacaine and 0.5mL of 10mg/mL dexamethasone on each side for total volume of 10 mL). Thirty minutes later and 24 hours following injection, the patient will rate their pain from 0-10 on the NRS. The description of the procedure is stated below. A success would be considered a drop in their pain score of at least 2.

Adverse effects will also be recorded 30 minutes after the procedure and the following day. Chart review on both provider and nursing notes will be performed on subsequent days to evaluate for adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Aneurysmal SAH in anterior/middle cerebral compartment
* Aneurysm must be secured endovascular with coiling
* The patient or patient's surrogate should be able to give informed consent and understand the risks of this study
* Pain NRS ≥ 5/10 in severity

Exclusion Criteria:

* Non aneurysmal, traumatic SAH
* Posterior fossa aneurysm ruptures
* Pregnancy
* Transcranial Doppler velocities suggestive of or approaching vasospasm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
Reduction in patient reported pain using a standard numeric rating scale (NRS) | 1 Day
  A combination of Bupivacaine 0.5% 4.5mL along with Dexamethasone 10mg/mL 0.5mL will be injected toward the sphenopalatine ganglion using a suprazygomatic approach bilaterally

CONTACTS AND LOCATIONS:
Overall Officials: Narayan Kissoon, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials